CLINICAL TRIAL: NCT03211546
Title: A Prospective Multicenter Observational Registry for Femoral Shaft Fractures in Children up to 16 Years of Age
Brief Title: Pediatric Femur Fracture Registry
Acronym: PedFemFx
Status: Completed | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: PedFemFx
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Femoral Shaft Fracture
Keywords: Pediatric femur fracture; Spica casting; Traction; Intramedullary nailing; Children; Internal fixation; External fixation
MeSH Terms: interventions — Therapeutics; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Femoral shaft fracture: Patients (children up to 16 years old) diagnosis of isolated closed femur shaft fracture (3.2-D) and open distal physis. Treatment strategies will follow standard of care (routine) procedures, either conservative (non-surgical) treatment or surgical treatment.
  Interventions: Procedure: Conservative (non-surgical) treatment; Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Conservative (non-surgical) treatment — Spica cast Traction Traction and spica cast
Procedure: Surgical treatment — Elastic Stable Intramedullary Nailing (ESIN) Conventional locking intramedullary nail Plating External fixation

SUMMARY:
Prospective data collection and evaluation of complete data sets will be performed in the course of routine clinical care of a cohort of consecutive patients (children up to 16 years old) presenting with an isolated femur shaft fracture. Data will be collected during follow-up visits at 3 to 6 weeks, 3, 6, 12 and 24 months, with additional follow-up visits as needed or dictated by individual practice. Final follow-up will be at 24 months, unless a patient requires additional follow-up or another intervention to address an unfavorable outcome (e.g. malalignment, nonunion, limb length discrepancy) noted at the 24 month follow-up visit.

DETAILED DESCRIPTION:
There is limited evidence about the comparative effectiveness of different treatments for pediatric femur fractures. The most common method used for isolated femur shaft fractures of children older than 5 years of age is elastic stable intramedullary nailing (ESIN). It is thought to be the ideal indication for children up to the age of 10 to 12 and it is the most commonly employed method of internal fixation in this age group, but other treatments include external fixation, plating, other forms of flexible or rigid intramedullary nailing and non-operative options such as spica casts or traction. In children under the age of 5 non-operative methods are believed to work well with few complications. Imperfect alignment is more acceptable because of the tremendous remodelling potential in young growing children. Internal fixation is believed to be unnecessary as it is more invasive, with some risk of complications and likely need for a second surgical procedure to remove it. Biomechanical properties are different in this age group. Consequently, operative treatment of these fractures is generally not recommended in children under the age of 3 according to the German guidelines (www.awmf.org), not under the age of 5 in the American guidelines (www.aaos.org); and in Great Britain, surgical management in preschool children is restricted to polytrauma and complex injuries (www.nice.org.uk).

Despite these recommendations and the general acceptance of non-operative treatment for younger children , a survey of clinical practice in Germany revealed that 50% of children under the age of 3 years are treated with ESIN, because some surgeons believe that patients seem less comfortable when treated with traction or spica casting and might experience a higher rate of loss of reduction. Consequently, the use of ESIN for fractures in preschool children has become more prevalent in the last years.

Similarly, there is wide variation in the preferred management of femoral shaft fractures in older children, with little evidence about the comparative effectiveness of different treatments for pediatric femur fractures. There is an imperative to collect prospective data to generate higher quality evidence.

The purpose of this proposed registry is to collect the clinical outcomes (fracture healing & patient reported outcomes and complications) of the treatment of isolated femur shaft fractures in children up to skeletal maturity. Additionally, health economic aspects will be evaluated to give possible recommendations from a health economic perspective.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 16 years of age at the time of the injury
* Open distal physis of the femur
* Diagnosis of isolated closed femur shaft fracture (3.2-D)
* Willingness and ability of the patient/parents/legally responsible care giver to participate in the clinical investigation including imaging and FU procedures as standard of care in each clinic
* Willingness and ability of the parent(s) to support the patient in his/her study participation
* Ability of parents to understand the content of the patient information / ICF and participation in the clinical investigation
* Signed ICF by patient and/or parent(s) according to local policies and regulations

Exclusion Criteria:

* Polytraumatized patient
* Closed distal physis of the femur
* Pathologic fractures and fractures in patients with metabolic bone disease, osteogenesis imperfecta, neuromuscular disorder, endocrinologic disease or other conditions influencing the bony structure
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Consecutive patients (children up to 16 years old) presenting with an isolated closed femur shaft fracture (3.2-D) and open distal physis.
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Fracture alignment | up to 24 months
  Mechanical and anatomical axes

SECONDARY OUTCOMES:
Range of Motion (ROM) | up to 24 months
  ROM of the hip (flexion/extension, internal/external rotation and abduction/adduction) and the knee (flexion/extension)
Axial deviation | up to 24 months
  Varus/valgus malalignment, flexion/extension deficit or rotational malalignment will be evaluated compared to the contralateral (healthy) leg
Leg Length Discrepancy | up to 24 months
  The Leg Length Discrepancy (LLD) will be measured using the standing blocks method
Quadriceps strength | up to 24 months
  The quadriceps strength will be measure using the manual muscle testing.
Return to full activity | up to 24 months
  ime to full weight-bearing, time to full activity, and time to return to kindergarten/school.
Patient-reported outcome | up to 24 months
  Patient Reported Outcomes of Fracture Healing- Lower Limb
Health Related Quality of Life | up to 24 months
  EQ-5D-Y version proxy 1

CONTACTS AND LOCATIONS:
Overall Officials: Peter P. Schmittenbecher, Prof., Principal Investigator — Kinderchirurgische Klinik, Klinikum Karlsruhe; Unni G. Narayanan, Prof., Principal Investigator — The Hospital for Sick Children, Toronto
Locations (14):
- Boston Children's Hospital, Boston, Massachusetts, United States
- Medical University Hospital of Graz, Graz, Austria
- Canada (4):
  - BC Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, New Scotland
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- Germany (6):
  - Universitätsklinik Dresden, Dresden
  - University Medicine Göttingen (UMG), Göttingen
  - Altonaer Kinderkrankenhaus GmbH, Hamburg
  - Städt. Klinikum Karlsruhe, Karlsruhe
  - University of Leipzig, Leipzig
  - University Hospital Tübingen, Tübingen
- Switzerland (2):
  - Inselspital, Bern
  - Childrens Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No